CLINICAL TRIAL: NCT04836117
Title: Evaluating the Impact of SomaSignal Tests on Medical Management and Change in Risk in Patients at Higher Risk of Cardiovascular Disease: A Feasibility and an Adaptive Implementation Study (SomaSignal Study)
Brief Title: Evaluating the Impact of SomaSignal Tests on Medical Management and Change in Risk in Patients at Higher Risk of Cardiovascular Disease: A Feasibility and an Adaptive Implementation Study
Acronym: SomaSignal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: SomaLogic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1051629
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Masking Description: All participants will know what group they are placed in. For Group 1 (Informed), clinicians and participants will receive their test results immediately. Those in Group 2 (Uninformed) will not receive their test results until study conclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informed (Experimental): Blood draw for SomaSignal Test and laboratory assessments at baseline, and 6 months (±30 days); SomaSignal Test results to be sent to investigators as available. Review and discussion of results with the participant from baseline and 6 months within 30 days (2-4 weeks to get SomaSignal results) after blood draw. Initiation of changes in medical management as soon as test results are known and discussed with patient.
  Patients will have a blood draw performed at baseline and 6 months for lipid panel, hemoglobin A1C, CBC, and BMP.
  Interventions: Other: SomaSignal Test Results
- Uninformed (No Intervention): Blood draw for SomaSignal Test at baseline and 6 months (+30 days). However, results will not be provided to clinician and participant until study conclusion. Patients contacted within 30 days (2-4 weeks) after baseline and 6-month visits to discuss treatment strategy (nothing, add/ remove medication, etc.) made at visit. Patients will have a blood draw performed at baseline and for lipid panel, hemoglobin A1C, CBC, and BMP
  SomaSignal Test results to be sent to investigators AFTER study conclusion. Patients will be provided with SomaSignal Test results after the 6 month post-test timepoint.

INTERVENTIONS:
Other: SomaSignal Test Results — SomaLogic, Inc. translates patterns from 5000 protein measurements made in thousands of participants in clinical trials into validated models (SomaSignal Tests) that predict important health outcomes or correlate with established health measures. SomaLogic, Inc. has developed these protein-based tests for the detection, subtyping and prognosis of heart disease and related medical, physiological and behavioral conditions. These tests are demonstrated in large retrospective studies to provide information superior to best available alternatives.
  Arms: Informed

SUMMARY:
Feasibility Study Informed consent will be obtained using an IRB-approved form. The first 12 consenting patients will be placed in the planned assessment group for feasibility and will not be randomized. These participants will undergo visits and blood draw collection at 3 months. They will be informed of their SomaSignal Test results at baseline and 3 months.

Recommendations for any medical management changes will be made based on an understanding of those results.

Randomized Study The succeeding 200 participants will be randomized using permuted mixed block randomization, in a 2:1 ratio, i.e., 2 participants to Group 1 (informed of their test results) and 1 participant to Group 2 (uninformed of their test results). At enrollment, and for 6 months thereafter, clinical information will be obtained from each participant's medical records, and/or directly from the participant during procedures, treatments, study-specific visits, and/or follow-up visits. Data collected for the study will have data linkage at SomaLogic, Inc., where data analysis will be done.

At baseline and 6-months (+30 days) post-enrollment, patients will undergo a patient visit and blood collection. Blood will be collected as a stand-alone sample collection, or when other ordered lab work is done, or from access lines inserted during a usual or specialized care. Samples will be sent to the Intermountain Central laboratory for clinical testing. A sample will also be processed and shipped to SomaLogic, Inc. for analysis at baseline and 6 months.

For the informed arm, the SomaSignal Test reports will be provided at the time they are available (2 to 4 weeks after the blood draw). Any recommended changes in medical management will be recorded in the case report forms and will be verified by the Principal Investigator.

For the uninformed arm, the SomaSignal Test results will not be provided to the study team until after the 6-month post-test visit. Adjustments, if any, would be made to the participant's management at that time.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 40 - 80 years of age
2. Receiving care at Intermountain Medical Center
3. At higher than typical risk for cardiovascular events, as assessed by the Principal Investigator or his/her delegate (further defined in the protocol)
4. Currently not pregnant
5. Ability to understand and sign a written informed consent form which must be obtained prior to initiation of any study procedures
6. Willing and able to comply with any virtual or in-person follow-up visits, tests, and schedule of evaluations
7. Willing and able to undergo a blood draw for SomaSignal Tests
8. Willing and able to provide access to their electronic health records

Exclusion Criteria:

1. Presence of Systemic Lupus Erythematosus
2. Inability to communicate appropriately
3. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study
4. Other conditions that in the opinion of the Principal Investigator and/or Co-Principal Investigators may increase risk to the participants and/or compromise the quality of the clinical trial
5. The Principal Investigator and/or Co-Principal Investigator determine(s) that the participant is not eligible for participation in this research study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-08-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Porportion of participants that undergo a change in their treatment plan after receipt of the SomaSignal test. | Baseline, 6 months
  Lifestyle changes are defined as referrals for
  * A structured dietary or weight loss program (ie., Intermountain's Weigh to Health)
  * Physical therapy for cardiovascular fitness
  * Cardiac rehabilitation Medications
  * Antianginals
  * Antiarrhythmics
  * Antilipidemics
  * Coagulation modifiers
  * Heart failure medications
  * Hypertension medications
  * Antidiabetic
  * Antiplatelets
  Patients will receive a point for each change made. Documentation will be made on whether the change was made because of the SomaSignal results, a side-effect or a request by the patient, or a non-SomaSignal test related reason. The total number of changes at baseline and 6-months will be computed for each patient and will be compared between the arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams SA, Murthy AC, DeLisle RK, Hyde C, Malarstig A, Ostroff R, Weiss SJ, Segal MR, Ganz P. Improving Assessment of Drug Safety Through Proteomics: Early Detection and Mechanistic Characterization of the Unforeseen Harmful Effects of Torcetrapib. Circulation. 2018 Mar 6;137(10):999-1010. doi: 10.1161/CIRCULATIONAHA.117.028213. Epub 2017 Oct 3. PMID 28974520
- [Background] Ganz P, Heidecker B, Hveem K, Jonasson C, Kato S, Segal MR, Sterling DG, Williams SA. Development and Validation of a Protein-Based Risk Score for Cardiovascular Outcomes Among Patients With Stable Coronary Heart Disease. JAMA. 2016 Jun 21;315(23):2532-41. doi: 10.1001/jama.2016.5951. PMID 27327800
- [Background] Williams SA, Kivimaki M, Langenberg C, Hingorani AD, Casas JP, Bouchard C, Jonasson C, Sarzynski MA, Shipley MJ, Alexander L, Ash J, Bauer T, Chadwick J, Datta G, DeLisle RK, Hagar Y, Hinterberg M, Ostroff R, Weiss S, Ganz P, Wareham NJ. Plasma protein patterns as comprehensive indicators of health. Nat Med. 2019 Dec;25(12):1851-1857. doi: 10.1038/s41591-019-0665-2. Epub 2019 Dec 2. PMID 31792462